CLINICAL TRIAL: NCT03015402
Title: Phase II Clinical Investigation of Oral Nitrite in Patients With Pulmonary Hypertension and Heart Failure With Preserved Ejection Fraction (PH-HFpEF)
Brief Title: Oral Nitrite in Patients With Pulmonary Hypertension and Heart Failure With Preserved Ejection Fraction
Acronym: PH-HFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Risbano, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY20010014; 5P01HL103455 (NIH)
Record Dates: First submitted 2017-01-05; First posted 2017-01-10 (Estimated); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Hypertension Secondary; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sodium Nitrite (Experimental): Study
  Interventions: Drug: Sodium Nitrite
- Placebo (Placebo Comparator): Control
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Sodium Nitrite — 40 mg PO (by mouth) TID (three times each day) for 10 weeks
  Other Names: study
  Arms: Sodium Nitrite
Drug: Placebo Oral Capsule — Placebo capsule that is of identical size, shape, and color to experimental drug capsule PO (by mouth) TID (three times each day) for 10 weeks
  Other Names: control
  Arms: Placebo

SUMMARY:
The main objective of this study is to determine the clinical efficacy of oral inorganic nitrite verses placebo and the therapeutic response with regards to exercise tolerance in patients with pulmonary hypertension and heart failure with preserved ejection fraction (PH-HFpEF).

DETAILED DESCRIPTION:
This is a single-center, 22-week double-blind, randomized placebo-controlled cross-over trial of oral nitrite on exercise capacity and hemodynamic measurements in subjects with PH-HFpEF.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years and older

PH-HFpEF confirmed diagnosis by RHC:

* Mean Pulmonary Arterial Pressure (mPAP) ≥ 25 mmHg AND
* Pulmonary capillary wedge pressure (PWCP) ≥ 15 mmHg AND
* Transpulmonary Gradient (TPG) ≥ 12 mmHg

Exclusion Criteria:

* Age less than 18 years;
* SBP > 170 or < 110 mmHg
* DBP >95 or < 60 mmHg
* Hemoglobin A1C > 10
* Positive urine pregnancy test or breastfeeding;
* Ejection Fraction (EF) < 40%;
* Dementia
* End-stage malignancy
* Major cardiovascular event or procedure within 6 weeks prior to enrollment
* Severe valvular disease
* Known chronic psychiatric or medical conditions that may increase the risk associated with study participation in the judgment of the investigator, would make the subject inappropriate for entry into this study;
* Smoker
* Hemoglobin <9 g/dL
* Serum creatinine > 3.0 mg/dL
* Receipt of an investigational product or device, or participation in a drug research study within a period of 15 days; RHC < 2 weeks from study screening RHC unless clinically indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Risbano, MD, MA, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 33 subjects were enrolled and consented with 9 screen failed/ineligible and 24 randomized. Of the 24 randomized, 3 were on drug/placebo but withdrew at a later time, and 21 completed the study.
Groups:
- Nitrite Then Placebo: Sodium Nitrite: 40 mg PO (by mouth) TID (three times each day) for 10 weeks, then crossover to receive placebo for 10 weeks.
- Placebo Then Nitrite: Placebo Oral Capsule: Placebo capsule that is of identical size, shape, and color to experimental drug capsule PO (by mouth) TID (three times each day) for 10 weeks, then crossover to receive nitrite for 10 weeks.
Period: First Intervention (10 Weeks)
Arm/Group | Nitrite Then Placebo | Placebo Then Nitrite
Started | 13 | 11
Completed | 13 | 9
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Washout (2 Weeks)
Arm/Group | Nitrite Then Placebo | Placebo Then Nitrite
Started | 13 | 9 (2 withdrew prior to the start of the washout period.)
Completed | 12 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention (10 Weeks)
Arm/Group | Nitrite Then Placebo | Placebo Then Nitrite
Started | 12 | 9
Completed | 12 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrite Then Placebo | Placebo Then Nitrite | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (7.0) | 69.6 (7.4) | 69.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24
Sitting Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 138 (17.4) | 131.5 (17.1) | 134.7 (17.2)
Sitting Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74.5 (9.8) | 75.9 (9.2) | 75.2 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: Mean Pulmonary Artery Pressure (mPAP) During Submaximal Exercise as Compared Between Placebo and Nitrite
Description: Mean Pulmonary Artery Pressure measurement at submaximal exercise as compared between Placebo and Oral Nitrite at 10 weeks.
Time Frame: Baseline and 10 weeks
Population: All participants who received at least one dose of each intervention and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Oral Nitrite: Participants who received Oral Nitrite in the first or last 10 weeks of the study.
- Placebo: Participants who received placebo in the first or last 10 weeks of the study.
Arm/Group | Oral Nitrite | Placebo
Number analyzed (Participants) | 21 | 21
mmHg
  Supine Mean Pulmonary Artery Pressure at Baseline | 48.75 (11.73) | 48.68 (11.34)
  Supine Mean Pulmonary Artery Pressure at 10 Weeks | 56.81 (9.87) | 55.0 (8.10)
Statistical Analysis 1: Comparison: Oral Nitrite vs Placebo; Test type: Superiority — Pre-randomization characteristics of 2 groups will be presented using the median (IQR) or frequency tables at each study sequence. The difference of mPAP during submax exercise compared between placebo and nitrite at 10 weeks (i.e. week 10 RHC of placebo vs week 10 RHC of nitrite) using parametric PK-cross analysis (i.e. ANOVA to determine the sequence, period, carryover, & treatment effects). Post-exercise values before & after crossover will be compared between 2 groups using similar approach; p = 0.20, ANOVA

2. Secondary Outcome: Difference in 6-minute Walk Test
Description: The 6-minute walk test measures the distance an individual is able to walk over 6 minutes on a hard, flat surface. The subject is allowed to self-pace and rest as needed.
  The number of subjects with available 6-minute walk tests do not match the total number of subjects in the study due to: one subject fracturing a foot and several subjects missing visit timepoints due to health issues resulting in 6 minute walk test not being performed.
Time Frame: Baseline to 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Oral Nitrite | Placebo
Number analyzed (Participants) | 19 | 19
meters
  Baseline Distance | 269.5 (130.3) | 253.2 (59.7)
  10 Weeks Distance | 267.6 (164.1) | 255.2 (89.3)

3. Secondary Outcome: Change in Right Heart Catheterization (RHC) Hemodynamics - Pulmonary Capillary Wedge Pressure
Description: Right heart catheterization hemodynamic measures will be aggregated to determine if overall hemodynamic on Pulmonary Capillary Wedge Pressure are improved over the course of treatment.
Time Frame: During Week 10 follow-up at rest and at exercise
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Nitrite | Placebo
Number analyzed (Participants) | 21 | 21
mmHg
  Pulmonary Capillary Wedge Pressure (Rest) | 28.2 (8.7) | 26.3 (7.9)
  Pulmonary Capillary Wedge Pressure (Exercise) | 29.9 (11.8) | 28.4 (10.5)

4. Secondary Outcome: Change in Severity of Heart Failure
Description: Determined by N-terminal pro b-type natriuretic peptide (NT-proBNP) plasma levels.
  The number of subjects with available NT-proBNP values do not match the total number in the study as several subjects missed visit timepoints due to health issues resulting in NT-proBNP not being obtained.
Time Frame: Baseline to Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oral Nitrite | Placebo
Number analyzed (Participants) | 19 | 19
pg/ml | 4146.055 (3357.261) | 4215.096 (3372.754)

5. Secondary Outcome: Change in Right Heart Catheterization (RHC) Hemodynamics - Trans Pulmonary Gradient
Description: Right heart catheterization hemodynamic measures will be aggregated to determine if overall hemodynamic on Trans Pulmonary Gradient are improved over the course of treatment.
Time Frame: During Week 10 follow-up at rest and at exercise
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Nitrite | Placebo
Number analyzed (Participants) | 21 | 21
mmHg
  Trans Pulmonary Gradient (Rest) | 20.6 (12.1) | 22.6 (11.1)
  Trans Pulmonary Gradient (Exercise) | 27.1 (11.2) | 26.6 (8.4)

6. Secondary Outcome: Change in Right Heart Catheterization (RHC) Hemodynamics - Pulmonary Vascular Resistance
Description: Right heart catheterization hemodynamic measures will be aggregated to determine if overall hemodynamic on Pulmonary Vascular Resistance are improved over the course of treatment.
Time Frame: During Week 10 follow-up at rest and at exercise
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Wood Units
Arm/Group | Oral Nitrite | Placebo
Number analyzed (Participants) | 21 | 21
Wood Units
  Pulmonary Vascular Resistance (Rest) | 3.2 (2.5) | 3.2 (2.5)
  Pulmonary Vascular Resistance (Exercise) | 3.4 (2.4) | 2.9 (1.5)

7. Secondary Outcome: Change in Right Heart Catheterization (RHC) Hemodynamics - Cardiac Output
Description: Right heart catheterization hemodynamic measures will be aggregated to determine if overall hemodynamic on Cardiac Output are improved over the course of treatment.
Time Frame: During Week 10 follow-up at rest and at exercise
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Oral Nitrite | Placebo
Number analyzed (Participants) | 21 | 21
liters per minute
  Cardiac Output (Rest) | 8.1 (2.4) | 8.8 (3.1)
  Cardiac Output (Exercise) | 9.4 (3.1) | 10 (3.1)

8. Secondary Outcome: Number of Participants With Different Severities of Heart Failure
Description: Determined by NYHA functional classification changes. Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  While the change in severity of heart failure is listed as an end point, since this is ordinal data we cannot provide a p-value. We present the NYHA data at screening, crossover and 10 weeks.
Time Frame: 10 weeks
Population: All participants who received at least one dose of each intervention and completed all study visits were included in the efficacy analysis.
  Not all subjects had NYHA Functional class assessed as some subjects missed appointments and some were lost due to the pandemic.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Nitrite | Placebo
Number analyzed (Participants) | 16 | 16
Participants
  Class I | 2 | 1
  Class II | 8 | 5
  Class III | 6 | 9
  Class IV | 0 | 1

9. Secondary Outcome: Change in Endurance Exercise Time
Description: The endurance exercise time will be measured from the start of loaded pedaling to volitional exhaustion and the worklaod has returned to unloaded pedaling.
Time Frame: 10 weeks
Population: All participants who received at least one dose of each intervention and completed all study visits were included in the efficacy analysis.
  This value represents the change in endurance time (difference in time measured while pedaling) from baseline to week 10 during cardiopulmonary exercise testing in minutes.
  Not all subjects had cardiopulmonary exercise testing performed due to missed visits related to personal health (i.e. fracture, or not feeling well to travel).
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Nitrite: Participants who received Oral Nitrite in the first or last 10 weeks of the study.
Arm/Group | Nitrite | Placebo
Number analyzed (Participants) | 18 | 18
minutes | -0.056 (2.526) | -0.904 (3.705)

ADVERSE EVENTS:
Time Frame: From Baseline through study completion, up to 26 weeks
Arm/Group | Oral Nitrite | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 22/24 | 23/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Nitrite (N=24) | Placebo (N=24)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (6) | 3 (3)
Heartburn (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hand,Food, and mouth (Infections and infestations) | 1 (1) | 0 (0)
Inflammation Right Ear (Infections and infestations) | 0 (0) | 1 (1)
Volume Overload (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 4 (4) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Chest Tightness (Cardiac disorders) | 4 (4) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Systolic Murmur (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness/Lightheadedness (Nervous system disorders) | 6 (6) | 8 (8)
Headache (Nervous system disorders) | 8 (8) | 5 (5)
Earache (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Inflammation of Ear (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vision Disturbance (Eye disorders) | 0 (0) | 1 (1)
Conjuctivitis (Eye disorders) | 0 (0) | 1 (1)
Influenza (General disorders) | 3 (3) | 2 (2)
Swelling of Extremity (General disorders) | 4 (4) | 5 (5)
Fatigue (General disorders) | 7 (7) | 7 (7)
Chills (General disorders) | 1 (1) | 0 (0)
SARS-CoV-2 Virus (General disorders) | 0 (0) | 1 (1)
Abscess of tooth (General disorders) | 1 (1) | 0 (0)
Cramps (General disorders) | 0 (0) | 1 (1)
Increased Potassium (General disorders) | 0 (0) | 1 (1)
Cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Gout Flare (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Increased Respiratory Rate (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bibasilar Crackles (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Stent Procedure (leg) (Vascular disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
This was a small clinical trial that under-enrolled due to the pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT03015402/Prot_SAP_000.pdf